CLINICAL TRIAL: NCT06726902
Title: Comparative Evaluation of the Effect of Different Adjunctive Air Polishing Powders in Nonsurgical Periodontal Therapy in Patients with Stage II and III Periodontitis: (A Randomized Controlled Clinical Trial)
Brief Title: Comparative Evaluation of the Effect of Different Adjunctive Air Polishing Powders in Nonsurgical Periodontal Therapy in Patients with Stage II and III Periodontitis
Acronym: GBT
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Diana Ibrahim (Other)
Responsible Party: Sponsor-Investigator, Diana Ibrahim, Periodontology MSc. Candidate, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IORG 0008839-0854-01/2024
Record Dates: First submitted 2024-12-06; First posted 2024-12-10 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Periodontitis
Keywords: GBT; Periodontitis; SI
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Test Group I (GBT and SI + erythritol powder) (Experimental): will receive GBT and SI with adjunctive air-polishing using Standard/ Subgingival nozzle + erythritol powder
  Interventions: Device: GBT and SI with erythritol powder
- Test Group II (GBT and SI + glycine powder) (Experimental): will receive GBT and SI with adjunctive air-polishing using Standard/ Subgingival nozzle + glycine powder
  Interventions: Other: GBT and SI with glycine powder
- Test Group III (GBT and SI + Trehalose powder) (Experimental): will receive GBT and SI with adjunctive air-polishing using Standard/ Subgingival nozzle + Trehalose powder
  Interventions: Other: GBT and SI with trehalose powder
- Control Group VI (SRP and SI) (Experimental): will receive conventional Scaling and Root planning (SRP) and (SI) without adjunctive air polishing powder
  Interventions: Other: SRP and SI

INTERVENTIONS:
Device: GBT and SI with erythritol powder — Non-Surgical Periodontal treatment:
  1. Guided Biofilm Therapy
     * Guided supragingival and shallow subgingival (PD ≥ 4 mm) removal of biofilm and stains from all quadrants using the air-polishing device using a standard nozzle system.
     * Subgingival removal of biofilm from deeper periodontal pockets (PD ≥ 6 mm) using an Air-polishing device subgingival nozzle system with erythritol powder .
  2. Scaling and root planing Scaling and root planing (SRP) For the control group, conventional scaling and root planning (SRP) only.
  Other Names: guided biofilm therapy
  Arms: Test Group I (GBT and SI + erythritol powder)
Other: GBT and SI with glycine powder — Non-Surgical Periodontal treatment:
  1. Guided Biofilm Therapy • Guided supragingival and shallow subgingival (PD ≥ 4 mm) removal of biofilm and stains from all quadrants using the air-polishing device using a standard nozzle system. • Subgingival removal of biofilm from deeper periodontal pockets (PD ≥ 6 mm) using an Air-polishing device subgingival nozzle system with glycine powder.
  2. Scaling and root planing Scaling and root planing (SRP) For the control group, conventional scaling and root planning (SRP) only
  Arms: Test Group II (GBT and SI + glycine powder)
Other: GBT and SI with trehalose powder — Non-Surgical Periodontal treatment:
  1. Guided Biofilm Therapy • Guided supragingival and shallow subgingival (PD ≥ 4 mm) removal of biofilm and stains from all quadrants using the air-polishing device using a standard nozzle system. • Subgingival removal of biofilm from deeper periodontal pockets (PD ≥ 6 mm) using an Air-polishing device subgingival nozzle system with trehalose powder .
  2. Scaling and root planing Scaling and root planing (SRP) For the control group, conventional scaling and root planning (SRP) only
  Arms: Test Group III (GBT and SI + Trehalose powder)
Other: SRP and SI — conventional scaling and root planning (SRP) with subgingival instrumentation only will be performed
  Arms: Control Group VI (SRP and SI)

SUMMARY:
The aim of this clinical trial is to evaluate and compare the effect of a newly designed air-polishing device (APD) using Erythritol, Glycine, and Trehalose air-polishing powders in nonsurgical periodontal therapy with control (conventional scaling and root planning) following the concept of guided biofilm therapy (GBT) as an adjunctive to subgingival instrumentation (SI) in nonsurgical periodontal therapy for Stage II and III periodontitis patients both clinically and microbiologically.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals of both sexes with an age between 30 and 65 years, having at least 16 natural teeth in function,
2. Stage II and III (moderate to severe) periodontitis, having at least 16 teeth with the need for SI
3. Interproximal plaque index (API) ≤ 35%; patients with Good oral hygiene.
4. No history of systemic disease that may influence periodontal disease

Exclusion Criteria:

1. Pregnancy or breastfeeding,
2. Smokers with more than seven cigarettes per day
3. Patients that had a treatment with antibiotics within six months before the study
4. Need for periodontal surgery or adjunctive antibiotic treatment to the SI
5. Patients who had any periodontal treatment during the last year before the study.
6. Patients with known systemic or autoimmune disease.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2024-03-03 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Bleeding on probing | up to six months
Pain Assessment | up to six months
  Pain level will be assed using Visual Analogue Scale (VAS) from 1 (minimum) to 10 (maximum)
Probing depth | up to six months
Plaque accumulation | up to six months
Clinical attachment level | up to six months
Microbiological Assessment of Aggregatibacter actinomycetemcomitans (Aa) | one month
Microbiological Assessment of Porphyromonas gingivalis (Pg) | one month
Microbiological Assessment of Tannerella forsythia (Tf) | one month
Microbiological Assessment of Treponema denticola (Td) | one month

CONTACTS AND LOCATIONS:
Overall Officials: Rania Abdelaziz Fahmy, PhD, Study Director — Alexandria University
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: six month